CLINICAL TRIAL: NCT00782327
Title: Randomized, Double-blind Study for the Evaluation of the Effect of Losartan Versus Placebo on Aortic Root Dilatation in Patients With Marfan Syndrome Under Treatment With Beta-blockers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008/503
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Marfan Syndrome
MeSH Terms: conditions — Marfan Syndrome | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Losartan
  Interventions: Drug: Losartan
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan — Daily maximal doses of Losartan will be 50mg for subjects under 50kg of weight and 100mg if the weight is over 50kg
  Arms: 1
Drug: Placebo — Daily placebo capsule
  Arms: 2

SUMMARY:
To study the effect of losartan (an angiotensin receptor blocker-ARB) on aortic root growth in patients with Marfan syndrome, already treated with beta-blockers (BB). The effect of losartan will be compared to placebo. Losartan or placebo will be added to the treatment regimen in a two-step up-titration scheme over 2 weeks. Start doses of Losartan will be 25 mg for subjects under 50kg of weight and 50mg if the weight is over 50kg. Uptitration will be guided by the tolerance of the drug by the patients. Patients will be contacted by phone call for assessment of side-effects before second step of uptitration.

Daily maximal doses of Losartan will be 50mg for subjects under 50kg of weight and 100mg if the weight is over 50kg

ELIGIBILITY:
Inclusion Criteria:

* Patients > 10 years
* Diagnosis of MFS, according to the Ghent criteria and/or genetically proven FBN1 mutations or linkage
* Consent obtained (written) either for the patient and for his/her parents (<18y
* Z-score of the aorta at the level of the sinus of Valsalva ≥2 (BSA adjusted)
* ARB naïve patients

Exclusion Criteria:

* Poor echocardiographic window,limiting the accurate measurement of the aortic root
* Contra-indication for ARB: Bilateral renal artery stenosis, renal function abnormalities (creatinine above normal for age), hyperkalemia
* Intolerance for ARB (eg angioedema)
* Pregnancy or breast feeding women
* Absence of effective contraception
* Liver function abnormalities
* Heart Failure
* Patients included in other clinical trial

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-11-01 (Actual); Primary Completion 2014-11-26 (Actual); Study Completion 2014-11-26 (Actual)

PRIMARY OUTCOMES:
The decrease of rate of aortic root growth measured by echocardiography at level of sinuses of Valsalva. The measure will be expressed in mm of growth per year and as Z-score. | At baseline and after 6 months, 1, 2 and 3 years follow-up

SECONDARY OUTCOMES:
Comparative arterial stiffness | At baseline and after 6 months, 1, 2 and 3 years follow-up
Evaluation of progression of aortic regurgitation | At baseline and after 6 months, 1, 2 and 3 years follow-up
Aortic dissection incidence | At baseline and after 6 months, 1, 2 and 3 years follow-up
Aortic root surgery | At baseline and after 6 months, 1, 2 and 3 years follow-up
Progression of mitral regurgitation | At baseline and after 6 months, 1, 2 and 3 years follow-up
Left ventricular size and function | At baseline and after 6 months, 1, 2 and 3 years follow-up
Skeletal and somatic traits | At baseline and after 6 months, 1, 2 and 3 years follow-up
Quality of life | At baseline and after 6 months, 1, 2 and 3 years follow-up
Genetic polymorphisms affecting clinical symptoms and response to treatment | End of study
Death | At baseline and after 6 months, 1, 2 and 3 years follow-up
Aortic stiffness as assessed by MRI | At baseline and after 1 year and 3 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Julie De Backer, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be